CLINICAL TRIAL: NCT00268645
Title: Open Trial of the Safety and Efficacy of Lantus for Insulin Naive Type 2 Diabetes Mellitus Patients or Patients Who Use Insulin Combined With 1 or More Oral Antidiabetic Drugs and Don't Have Good Glycemic Control.
Brief Title: Insulin Glargine in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_5036
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine

SUMMARY:
The aim of this project is to confirm the efficacy and safety profile of Insulin glargine in daily practice and to improve the physicians' knowledge and experience concerning Insulin glargine

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus patients,
* Diabetic patients receiving insulin or patients who are insulin-naive and whose glycemic control cannot be sufficiently maintained with single or combined oral antidiabetic agents,
* Patients with HbA1C>8
* Patients able to self-measure its blood glucose levels.

Exclusion Criteria:

* According to package insert information (Summary of Product Characteristics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534
Dates: Start 2004-09

PRIMARY OUTCOMES:
For efficacy: FBG (Fasting Blood Glucose), HbA1c

SECONDARY OUTCOMES:
For safety: ICA (Insulin Cell Antibody)

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)